CLINICAL TRIAL: NCT00781664
Title: 21-Day Cumulative Irritation Test
Brief Title: Cumulative Irritation Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AN2718-TP-101
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — Sodium Dodecyl Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- A (Experimental): AN2718 Cream SF Vehicle
  Interventions: Other: AN2718
- B (Experimental): AN2718 Cream SF, 0.3%
  Interventions: Drug: AN2718
- C (Experimental): AN2718 Cream SF, 1%
  Interventions: Drug: AN2718
- D (Experimental): AN2718 Gel Vehicle
  Interventions: Other: AN2718
- E (Experimental): AN2718 Gel, 1.5%
  Interventions: Drug: AN2718
- F (Experimental): AN2718 Gel, 2.5%
  Interventions: Drug: AN2718
- G (Experimental): AN2718 Gel, 5%
  Interventions: Drug: AN2718
- H (Experimental): AN2718 Gel, 7.5%
  Interventions: Drug: AN2718
- I (Active Comparator): Sodium Lauryl Sulfate, 0.5%
  Interventions: Other: Sodium Lauryl Sulfate

INTERVENTIONS:
Other: AN2718 — AN2718 Cream SF Vehicle, Daily for up to 21 days
  Arms: A
Drug: AN2718 — AN2718 Cream SF, 0.3%, Daily for up to 21 days
  Arms: B
Drug: AN2718 — AN2718 Cream SF, 1%, Daily for up to 21 days
  Arms: C
Other: AN2718 — AN2718 Gel Vehicle, Daily for up to 21 days
  Arms: D
Drug: AN2718 — AN2718 Gel, 1.5%, Daily for up to 21 days
  Arms: E
Drug: AN2718 — AN2718 Gel, 2.5%, Daily for up to 21 days
  Arms: F
Drug: AN2718 — AN2718 Gel, 5%, Daily for up to 21 days
  Arms: G
Drug: AN2718 — AN2718 Gel, 7.5%, Daily for up to 21 days
  Arms: H
Other: Sodium Lauryl Sulfate — Sodium Lauryl Sulfate, 0.5%, Daily for up to 21 days
  Other Names: SLS
  Arms: I

SUMMARY:
The purpose of this study is to determine the cumulative irritation potential of the products listed by the Sponsor.

DETAILED DESCRIPTION:
Healthy, adult volunteers of either sex will be patched daily on his/her back with multiple strengths of AN2718 in 2 different topical dosage forms and an active comparator over the course of 21 consecutive days. Twenty-four hours after each application, the patches will be removed and the site evaluated using a five-point scale for irritation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria for inclusion in the study.

1. Healthy volunteers of either sex, at least 18 years of age or older.
2. Females must be of non-childbearing potential (i.e., post-menopausal or surgically sterile [bilateral oophorectomy and/or total hysterectomy]). All females must submit to a urine pregnancy test and have a negative result at Day 1 and at the final study visit.
3. Subjects may be of any skin type or race providing their degree of skin pigmentation does not interfere with making readings of skin reactions.
4. Willingness to follow the study procedures and complete the study.
5. Written informed consent obtained.

Exclusion Criteria:

1. Any skin disease that would in any way confound interpretation of the study results. Atopic dermatitis/eczema, psoriasis will be excluded.
2. Chronic asthma will be excluded.
3. Pregnant or nursing mothers.
4. A history of sensitivity to any component of any of the formulations.
5. Use of chronic medications (such as antihistamines, corticosteroids, analgesics and anti-inflammatories) for one week before and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Irritation Score (5-point scale) | Daily for 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- The Education and Research Foundation, Inc., Lynchburg, Virginia, United States